CLINICAL TRIAL: NCT03410147
Title: A Dose-finding and Feasibility Study for a Prolonged 13C-octanoate Breath Test for Gastric Emptying During Continuous Nutrient Infusion
Brief Title: A Dose-finding and Feasibility Study for a Prolonged 13C-octanoate Breath Test for Gastric Emptying
Acronym: ANTERO-AC-7
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, prof. dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: S61107
Record Dates: First submitted 2018-01-18; First posted 2018-01-25 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Healthy; Gastric Emptying
MeSH Terms: interventions — Gastric Emptying

STUDY DESIGN:
Intervention Model Description: A single blind, randomized, crossover monocentric study in a cohort of adult healthy volunteers
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Concentration A (Other): Concentration of 13C-sodium octanoate in enteral nutrition is 0.3 mg/ml
  Interventions: Diagnostic Test: 13C-octanoate breath test for gastric emptying
- Concentration B (Other): Concentration of 13C-sodium octanoate in enteral nutrition is 1.0 mg/ml
  Interventions: Diagnostic Test: 13C-octanoate breath test for gastric emptying
- Concentration C (Other): Concentration of 13C-sodium octanoate in enteral nutrition is 3.0 mg/ml
  Interventions: Diagnostic Test: 13C-octanoate breath test for gastric emptying

INTERVENTIONS:
Diagnostic Test: 13C-octanoate breath test for gastric emptying — The 13C-octanoate breath test for gastric emptying will be performed to assess gastric emptying rate of a liquid meal that is infused continuously over a period of 8 hour.
  13C-labeled sodium octanoate (food adjective) is mixed with liquid nutrients used for enteral feeding. The concentration of 13C-labeled sodium octanoate is according to the randomized treatment order. This mixture is infused at 20 ml/h for 8 hours (hourly dose of 13C-octanoate differs between treatment arms). In order to estimate gastric emptying rate quantitatively throughout the infusion period, the appearance of 13CO2 in the breath, relative to 12CO2, will be monitored by sampling the exhaled breath at a 15 minute interval.
  The aim is to induce a steady state hourly 13C-recovery. This would allow to implement the prolonged breath test protocol in future clinical investigations.

SUMMARY:
The objective of this dose-finding and feasibility study is to establish the optimal 13C-octanoate concentration to be used with slowly infused enteral nutrition to perform a prolonged gastric emptying test using the breath test. More specifically, the aim is to discover the 13C-octanoate concentration that induces a steady state hourly 13C-recovery. This would allow to implement the prolonged breath test protocol in a future clinical investigation in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* At least 18 years old
* BMI between and including 18 and 29
* Understand and able to read Dutch
* In good health on the basis of medical history
* Refrains from herbal, vitamin and other dietary supplements on the day of the visits

Exclusion Criteria:

* Dyspeptic symptoms (assessed with PAGI-SYM questionnaire, Annex II)
* Using any medication that might affect gastric function or visceral sensitivity
* Known / suspected current use of illicit drugs
* Known psychiatric or neurological illness
* Any gastrointestinal surgery that could influence normal gastric function in the opinion of the investigator
* History of heart or vascular diseases like irregular heartbeats, angina or heart attack
* Nasopharyngeal surgery in the last 30 days
* Suspected basal skull fracture or severe maxillofacial trauma
* History of thermal or chemical injury to upper respiratory tract or esophagus
* Current esophageal or nasopharyngeal obstruction
* Known coagulopathy
* Known esophageal varices
* Have a known allergy or intolerance to cow milk, soy or any other ingredient of Isosource Standard.
* Known galactosaemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Hourly 13C-recovery | 8 hour
  Indicator for gastric emptying rate

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium